CLINICAL TRIAL: NCT06480643
Title: Effect of Exercise Type on Muscle Quality in Patients With OA, SARC and RA: an Explorative Study The Care for Muscle Study
Brief Title: Effect of Exercise Type on Muscle Quality in Patients With OA, SARC and RA: an Explorative Study
Acronym: C4M
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Amsterdam UMC, location VUmc (Other)
Responsible Party: Principal Investigator, Maia Sobejana, Head researcher, Amsterdam UMC, location VUmc
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 86908
Record Dates: First submitted 2024-06-17; First posted 2024-06-28 (Actual); Last update posted 2024-06-28 (Actual); Status verified 2024-06

CONDITIONS: Rheumatoid Arthritis; Osteoarthritis; Sarcopenia
Keywords: exercise therapy; RMD; strength training; muscle endurance; rheumatoid arthritis; osteoarthritis; sarcopenia
MeSH Terms: conditions — Arthritis, Rheumatoid; Osteoarthritis; Sarcopenia

STUDY DESIGN:
Intervention Model Description: two-arm parallel-group exploratory trial including a total of 69 patients
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High load exercise type (Experimental): The patients will perform 6-8 full-body exercises using a load of 60-75% of their 1RM. The exercises will comprise of both compound (multi-joint movement that works multiple muscle groups at the same time) and isolation (movement that targets a single muscle group and involves the movement of a single joint) exercises. Each training session will be preceded by a 3-5mins warm-up. Total exercise duration will vary between 45-60mins, comprising of 3 sets of 10 repetitions with 1 min periods of recovery. Patients will be required to maintain an intensity of 7-8 on a 10-point physical exertion scale
  Interventions: Other: High load exercise type
- Low load exercise type (Experimental): Patients will perform 6-8 full-body exercises with a load of 30-45% of their 1RM. This training session will include both bodyweight and circuit training types. Each training session will be preceded by a 5-10mins warm-up. Total exercise duration will vary between 45-60mins (including the warm-up and cool down), with each exercise comprising of 3 sets of 20 repetitions with 1 min periods of recovery. A 5-min cool-down will follow the final rest period. Patients will be required to maintain an intensity of 7-8 on a 10-point physical exertion scale
  Interventions: Behavioral: Low load exercise type

INTERVENTIONS:
Other: High load exercise type — Heavier load, fewer reps
  Arms: High load exercise type
Behavioral: Low load exercise type — Lighter load, more reps
  Arms: Low load exercise type

SUMMARY:
C4M hypothesizes that patients with low muscle strength may respond differently to different types of exercise intervention, dependent on the underlying aetiology, i.e. impaired protein synthesis versus metabolic dysfunction and that this response is predictable based on the clinical diagnosis, i.e. rheumatoid arthritis (RA), osteoarthritis (OA) and Sarcopenia alone (SARC) and a number of clinical, blood based and muscle metabolic and architectural biomarkers. Understanding the underlying biochemical response of each patient group to the different type of exercise loading could help with the development of disease-specific training, making it more effective and more predictable on outcomes.

DETAILED DESCRIPTION:
Rationale: C4M hypothesizes that patients with low muscle strength may respond differently to different types of exercise intervention, dependent on the underlying aetiology, i.e. impaired protein synthesis versus metabolic dysfunction and that this response is predictable based on the clinical diagnosis, i.e. rheumatoid arthritis (RA), osteoarthritis (OA) and Sarcopenia alone (SARC) and a number of clinical, blood based and muscle metabolic and architectural biomarkers. Understanding the underlying biochemical response of each patient group to the different type of exercise loading could help with the development of disease-specific training, making it more effective and more predictable on outcomes.

Objective: to explore effectivity, interaction and predictability of two types of exercise intervention in patients with RA, OA and SARC alone. The primary outcome of this study will be isokinetic muscle strength of the quadriceps in all three target groups.

Study design: two-arm parallel-group exploratory trial including a total of 69 patients: study population 23 patients with OA, 23 patients with RA and 23 patients with SARC alone (according to the revised European Working Group on Sarcopenia in Older People consensus definition (EWGSOP-II criteria, Cruz- Jentoft 2019).

Intervention: Exercise intervention for 3 times a week for 8 weeks.

Main study parameters/endpoints: the main study parameter is the difference in isokinetic muscle strength pre- and post-intervention in all three patient groups. The secondary study parameters include muscle endurance; mitochondrial respiration, gene and protein expression and histology via muscle biopsies; inflammation via bloodwork and feasibility.

Intervention: Exercise intervention for 3 times a week for 8 weeks.

Main study parameters/endpoints: the main study parameter is the difference in isokinetic muscle strength pre- and post-intervention in all three patient groups. The secondary study parameters include muscle endurance; mitochondrial respiration, gene and protein expression and histology via muscle biopsies; inflammation via bloodwork and feasibility.

ELIGIBILITY:
Inclusion Criteria For all patients

* Low muscle strength defined as hand grip strength (HGS) <27 kg and <16 kg for males and females respectively. If HGS is not possible due to interfering pain or joint- deformity, the chair stand test is used instead, with low muscle strength defined as not able to rise from the chair without arms or a time >15 sec (Cruz Jentoft 2019).
* Gait speed of >0.8m/s to exclude patients who are too disabled to participate in the study (Cruz Jentoft 2019).

OA patients

* Age between 50 and 70
* Patients with either knee and/or hip OA according to clinical American College of Rheumatology (ACR) criteria (Altman 1986).
* Kellgren and Lawrence grading score of 2-4 for hip and/or knee OA (Altman 1991).
* C-reactive Protein (CRP) levels <10mg/L within 3 months prior to enrolment (Sanchez 2014).

Rheumatoid arthritis patients

* Age between 50 and 70
* Diagnosed with RA according to European Alliance of Associations for Rheumatology (EULAR)/ACR criteria (Aletaha 2010).
* Disease activity score in 28 joints (DAS28) 2.8<5.6, as defined by the EULAR criteria (Aletaha 2010), either de novo or despite Disease-Modifying Antirheumatic Drug therapy.
* Stable disease three months prior to the start of the exercise intervention.
* Stable rheumatic medication three months prior to the start of the exercise intervention.
* Stopped the usage of corticosteroids 3 months prior to the start of the exercise intervention.
* Disease duration >1 year and <15 years

Sarcopenia patients

* Age between 50 and 80.
* Sarcopenia without joint involvement (no OA, RA), according to the EWGSOPII criteria (Cruz Jentoft 2019) of low muscle strength defined as HGS <27kg and <16 kg for males and females respectively (dynapenia). This group will therefore primarily involve participants with probable sarcopenia (dynapenia) but may also encompass participants with confirmed sarcopenia (appendicular muscle Lean Mass (ALM)/height2 <7.0 kg/m2 for males and <5.5 kg/m2 for females) as this is not a selection criterion. Severe sarcopenia will be excluded (gait speed <0,8 m/s).
* Exclude patients with joint complaints (RA, OA, or other joint disease).

Exclusion Criteria:

* Body mass index (BMI) < 18 and > 35 Kg/m2
* Contra-indications for exercise testing and prescription as indicated by the ACSM guideline (i.e. progressive increase in heart failure symptoms, myocardial infarction less than three months before the start of the training programme, severe cardiac ischemia upon exertion, respiratory frequency of more than 30 breaths per minute and heart rate at rest >110 beats per minute).
* Participants taking beta-blockers for the duration of the intervention.
* Diagnosed with other neurologic or cachectic diseases or major surgery that may interfere with muscle quality (i.e. multiple sclerosis, ongoing cancer treatment or radiotherapy/ chemotherapy in the previous 6 months).
* Participating in another regular and intense (i.e. high physical loading training such as high-load circuit training for muscle gain and fat loss > 2 times a week) physical training programme within 2 months prior to enrolment.
* Ligament/muscle tear and/or other injuries within 6 months.
* Taking drugs (e.g. performance enhancing drugs) or nutritional supplements (e.g. protein powder) known to increase muscle mass.
* Inability to be scheduled for exercise therapy
* Insufficient comprehension of Dutch language or no informed consent.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
Isokinetic muscle strength in Nm/kg | Measured before and after the 8 week- exercise block.
  Maximal net joint moment measurements of muscle strength will be assessed using an isokinetic dynamometer (EnKnee, Enraf-Nonius, Rotterdam, the Netherlands). An initial practice attempt will be used for familiarization. Participants will perform three maximal test repetitions to measure the isokinetic strength of the quadriceps and hamstrings for each knee, at 60°/s. Mean quadriceps and hamstring muscle strength per leg will be calculated (in Nm) and divided by the participant's weight (in kg). Muscle strength data (in Nm/kg) of the index knee (most affected knee) will be used (de Zwart 2022). The 1-RM will be defined as the maximal weight in kg a patient could lift for only one repetition

SECONDARY OUTCOMES:
Muscle endurance in number of repetitions | Measured before and after the 8 week- exercise block.
  this will be measured by the knee extension test of both legs using an isokinetic dynamometer (EnKnee, Enraf-Nonius, Rotterdam, the Netherlands). The patients will be asked to perform the knee extension exercise at 30% 1RM until muscular failure. The number of repetitions obtained until muscular failure will be the indication of muscle endurance.
Myogenesis | Measured before the 8 week- exercise block.
  SETD3; MYOD1; MYOG
Apoptosis & proteolysis | Measured before the 8 week- exercise block.
  CASP1; CASP3; MURF1; MAFBX; BCL2; Gene + protein USP19
Oxidative stress & endogenous antioxidants | Measured before the 8 week- exercise block.
  3NT, Cys-S-NO, MDA*, NOS, NOX, GTHP, GTHO & SOD2; SOD1; CAT; HMOX1; NQO1; NRF2; GPX1
Mitochondrial biogenesis & function | Measured before the 8 week- exercise block.
  PPARGC1A; mitochondrial complex I-V (Ci-Cv); NDUFA1, NDUFA2, SDHA, SHDB, UQCRC1, CYC1, COX4I1, COX5A, ATP5B, ATP5A1, CCO, C15ORF48
Glucose metabolism | Measured before the 8 week- exercise block.
  GLUT4; SIRT1; FOXO1; AMPK-P
General inflammatory markers | Measured before and after the 8 week- exercise block.
  CRP, ESR
Cytokines | Measured before and after the 8 week- exercise block
  TNFa; IL1b; IL6; IFNy & myokines

OTHER OUTCOMES:
Age in years | Measured before 8 week- exercise block.
  Subject characteristic
Gender (male or female) | Measured before 8 week- exercise block.
  Subject characteristic
Height in centimetres | Measured before and after the 8 week- exercise block.
  Subject characteristic
Weight in kilgorams | Measured before and after the 8 week- exercise block.
  Subject characteristic
Co-morbidities | Measured before 8 week- exercise block.
  If any is present
Medication | Measured before 8 week- exercise block.
  Any current medication use or medication use in the past 3-6 months will be recorded.
Educational level | Measured before 8 week- exercise block.
  Highest level of education received
Employment status | Measured before 8 week- exercise block.
  Employed or unemployed
Marital status | Measured before 8 week- exercise block.
  Single, married, divorce, widow etc.
Smoking use | Measured before 8 week- exercise block.
  Smoking yes or no
Smoking frequency per day | Measured before and after the 8 week- exercise block.
  If patients smoke, the amount of cigarettes per day
Alcohol frequency | Measured before and after the 8 week- exercise block.
  If patients drink, the frequency in a day/week
Alcohol use | Measured before and after the 8 week- exercise block.
  Alcohol yes or no
BMI in kg/m^2 | Measured before and after the 8 week- exercise block.
  Anthropometric
Absolute & relative muscle mass in kilograms | Measured before and after the 8 week- exercise block.
  InBody S10, Biospace Co., Ltd, Seoul, South Korea) will be used to measure muscle mass. DSM-BIA has been validated for assessing segmental and whole-body composition against dual energy X-ray absorptiometry (DEXA) (Ling 2011). DSM-BIA will not be performed in patients with 1) electronic internal medical devices or implants such as cardiac pacemakers; 2) plasters or bandages interfering with the placement of the electrodes; 3) amputation.
Short-form mini-nutritional assessment | Measured before and after the 8 week- exercise block.
  Anthropometrics
Handgrip strength in kilograms | Measured before and after the 8 week- exercise block.
  A hand-held dynamometer (JAMAR, Sammons Preston, Inc., 119 Bolingbrook, IL, USA will be used to measure handgrip strength. Subjects will be in a sitting position with elbows flexed at 90 degrees, shoulders adducted and forearms in a neutral position without support and instructed to squeeze the dynamometer maximally three times for each hand, alternating between the right and the left- hand side. Maximal value will be reported in kg.
Short physical performance battery test (score 0-12) | Measured before and after the 8 week- exercise block.
  The total score of the SPPB is the sum of the number of points achieved (range between 0 and 12) in each of the test components. The higher the score, the better the patient's performance. Persons with a score between 4 and 9 have an increased risk of new disabilities and are therefore a suitable target group for interventions to improve functioning. People with a higher score are not yet in the danger zone. People with a lower score already experience many limitations and are therefore more likely to be eligible for interventions to maintain functioning and possibly deal with limitations.
6 minutes walk test in metres | Measured before and after the 8 week- exercise block.
  The 6 Minute Walk Test is a sub-maximal exercise test used to assess aerobic capacity and endurance. The distance covered over a time of 6 minutes is used as the outcome by which to compare changes in performance capacity.
FitMáx© survey in score | Measured before and after the 8 week- exercise block.
  The FitMáx© is a questionnaire consisting of three single answer questions, about the maximum capacity of walking, climbing stairs and cycling. The questionnaire consists of a scale from 0-13 to rate maximum capacity of walking, a scale from 0-11 for maximum capacity of cycling and for the maximum capacity of stair climbing a scale from 0-10 is used.
Patient-Reported Outcome Measures (PROMs) | Measured before and after the 8 week- exercise block.
  PROMIS-CAT short forms will be used to self-report of core symptoms and health-related quality of life according to the Item Response Theory. We will assess the domains pain, fatigue, physical function, social function (Witter 2016)
Muscle volume in m^2 | Measured before and after the 8 week- exercise block.
  Muscle volume will be measured between the origin and distal end of the muscle belly using manual segmentation of the anatomical cross-sections and interpolation in custom software. Average fascicle length (ℓfasc) and pennation angles (αfasc) will be estimated.
Average fascicle length (ℓfasc) | Measured before and after the 8 week- exercise block.
  Muscle volume will be measured between the origin and distal end of the muscle belly using manual segmentation of the anatomical cross-sections and interpolation in custom software. Average fascicle length (ℓfasc) and pennation angles (αfasc) will be estimated.
Pennation angles (αfasc) | Measured before and after the 8 week- exercise block.
  Muscle volume will be measured between the origin and distal end of the muscle belly using manual segmentation of the anatomical cross-sections and interpolation in custom software. Average fascicle length (ℓfasc) and pennation angles (αfasc) will be estimated.
Muscle physiological cross-sectional area (PCSA) | Measured before and after the 8 week- exercise block.
  PCSA will be calculated by dividing muscle volume by ℓfasc. Muscle volume and PCSA will are prime determinants of maximal muscle power and muscle strength, respectively.

REFERENCES:
- [Background] Dardevet D, Remond D, Peyron MA, Papet I, Savary-Auzeloux I, Mosoni L. Muscle wasting and resistance of muscle anabolism: the "anabolic threshold concept" for adapted nutritional strategies during sarcopenia. ScientificWorldJournal. 2012;2012:269531. doi: 10.1100/2012/269531. Epub 2012 Dec 23. PMID 23326214
- [Background] Bao W, Sun Y, Zhang T, Zou L, Wu X, Wang D, Chen Z. Exercise Programs for Muscle Mass, Muscle Strength and Physical Performance in Older Adults with Sarcopenia: A Systematic Review and Meta-Analysis. Aging Dis. 2020 Jul 23;11(4):863-873. doi: 10.14336/AD.2019.1012. eCollection 2020 Jul. PMID 32765951
- [Background] Ganz DA, Latham NK. Prevention of Falls in Community-Dwelling Older Adults. N Engl J Med. 2020 Feb 20;382(8):734-743. doi: 10.1056/NEJMcp1903252. No abstract available. PMID 32074420
- [Background] Hunter DJ, Bierma-Zeinstra S. Osteoarthritis. Lancet. 2019 Apr 27;393(10182):1745-1759. doi: 10.1016/S0140-6736(19)30417-9. PMID 31034380
- [Background] Hanaoka BY, Ithurburn MP, Rigsbee CA, Bridges SL Jr, Moellering DR, Gower B, Bamman M. Chronic Inflammation in Rheumatoid Arthritis and Mediators of Skeletal Muscle Pathology and Physical Impairment: A Review. Arthritis Care Res (Hoboken). 2019 Feb;71(2):173-177. doi: 10.1002/acr.23775. Epub 2019 Jan 4. PMID 30295435
- [Background] van Vilsteren M, Boot CR, Knol DL, van Schaardenburg D, Voskuyl AE, Steenbeek R, Anema JR. Productivity at work and quality of life in patients with rheumatoid arthritis. BMC Musculoskelet Disord. 2015 May 6;16:107. doi: 10.1186/s12891-015-0562-x. PMID 25940578
- [Background] Chen L, Nelson DR, Zhao Y, Cui Z, Johnston JA. Relationship between muscle mass and muscle strength, and the impact of comorbidities: a population-based, cross-sectional study of older adults in the United States. BMC Geriatr. 2013 Jul 16;13:74. doi: 10.1186/1471-2318-13-74. PMID 23865675
- [Background] Mayhew AJ, Amog K, Phillips S, Parise G, McNicholas PD, de Souza RJ, Thabane L, Raina P. The prevalence of sarcopenia in community-dwelling older adults, an exploration of differences between studies and within definitions: a systematic review and meta-analyses. Age Ageing. 2019 Jan 1;48(1):48-56. doi: 10.1093/ageing/afy106. PMID 30052707
- [Background] Helliwell PS, Jackson S. Relationship between weakness and muscle wasting in rheumatoid arthritis. Ann Rheum Dis. 1994 Nov;53(11):726-8. doi: 10.1136/ard.53.11.726. PMID 7826134
- [Background] Lemmey AB, Wilkinson TJ, Clayton RJ, Sheikh F, Whale J, Jones HS, Ahmad YA, Chitale S, Jones JG, Maddison PJ, O'Brien TD. Tight control of disease activity fails to improve body composition or physical function in rheumatoid arthritis patients. Rheumatology (Oxford). 2016 Oct;55(10):1736-45. doi: 10.1093/rheumatology/kew243. Epub 2016 Jun 10. PMID 27288209
- [Background] Steinz MM, Persson M, Aresh B, Olsson K, Cheng AJ, Ahlstrand E, Lilja M, Lundberg TR, Rullman E, Moller KA, Sandor K, Ajeganova S, Yamada T, Beard N, Karlsson BC, Tavi P, Kenne E, Svensson CI, Rassier DE, Karlsson R, Friedman R, Gustafsson T, Lanner JT. Oxidative hotspots on actin promote skeletal muscle weakness in rheumatoid arthritis. JCI Insight. 2019 Mar 28;5(9):e126347. doi: 10.1172/jci.insight.126347. PMID 30920392